CLINICAL TRIAL: NCT03039660
Title: Evidence-Based Online Curriculum to Improve Sleep in Medical Students: A Multisite Trial to Assess Efficacy and Feasibility of RefreshMD
Brief Title: Feasibility and Efficacy Study of Student Wellness Online Course for Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sara Grace Connolly, Medical Student, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RefreshMD
Record Dates: First submitted 2017-01-27; First posted 2017-02-01 (Estimated); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Student Wellness

ARMS (2):
- RefreshMD (Experimental): An online course for sleep improvement in medical students
  Interventions: Behavioral: RefreshMD
- Bond Between Us (Placebo Comparator): An online course covering communication skills and the physician-patient relationship
  Interventions: Behavioral: Bond Between Us

INTERVENTIONS:
Behavioral: RefreshMD — Online Sleep Improvement Course
  Arms: RefreshMD
Behavioral: Bond Between Us — Online Educational Course
  Arms: Bond Between Us

SUMMARY:
This study aims to investigate the feasibility and efficacy of online student wellness courses for improving medical student mental health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Full-time medical student at a participating medical school
* Will remain enrolled as full-time medical student throughout duration of study

Exclusion Criteria:

* Not a full-time medical student at a participating medical school

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Enrollment numbers per course | 2 weeks
  # of participants who enroll / # of participants invited to enroll
Views per video | Throughout the course (6 weeks)
Number of actively engaged students per course | Throughout the course (6 weeks)

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Related Impairment | Through study completion (4 months)
PROMIS Sleep Disturbance | Through study completion (4 months)
PROMIS Depression | Through study completion (4 months)
Stanford Medical Student Burnout Questionnaire | Through study completion (4 months)

CONTACTS AND LOCATIONS:
Overall Officials: Sara G Cadman, MD, Principal Investigator — Stanford University graduate, Penn Medicine Fellow
Locations (3):
- United States (3):
  - Stanford University, Stanford, California
  - Washington University in St Louis, St Louis, Missouri
  - Rutgers Robert Wood Johnson, Piscataway, New Jersey